CLINICAL TRIAL: NCT01623375
Title: A Trial Investigating the Absolute Bioavailability of Insulin Degludec in Healthy Subjects
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Novo Nordisk A/S (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: NN1250-4000; 2012-000078-50 (EudraCT Number); U1111-1126-8860 (Other: WHO)
Record Dates: First submitted 2012-06-04; First posted 2012-06-20 (Estimated); Last update posted 2015-02-19 (Estimated); Status verified 2015-02

CONDITIONS: Diabetes; Healthy
MeSH Terms: conditions — Diabetes Mellitus | interventions — insulin degludec

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- s.c. (Experimental)
  Interventions: Drug: insulin degludec
- i.v. (Experimental)
  Interventions: Drug: insulin degludec

INTERVENTIONS:
Drug: insulin degludec — A single dose of 0.4 U/kg body weight will be administered subcutaneously (s.c., under the skin).
  Arms: s.c.
Drug: insulin degludec — A single dose of 0.04 U/kg body weight will be administered intravenously (i.v., into the vein).
  Other Names: IDeg
  Arms: i.v.

SUMMARY:
This trial is conducted in Europe. The aim of the trial is to investigate the absolute bioavailability of insulin degludec (IDeg) in healthy subjects.

ELIGIBILITY:
Inclusion Criteria:

* Considered generally healthy upon completion of medical history, physical examination, analysis of laboratory safety variables, vital signs and ECG (electrocardiogram), as judged by the investigator
* Body mass index 18.0-27.0 kg/m^2 (both inclusive)

Exclusion Criteria:

* Subject who has donated any blood or plasma in the past month or more than 500 mL within 3 months prior to screening
* Smoker (defined as a subject who is smoking more than 5 cigarettes or the equivalent per day)
* Not able or willing to refrain from smoking and use of nicotine gum or transdermal nicotine patches during the inpatient period

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 18 (Actual)
Dates: Start 2012-06; Primary Completion 2012-08 (Actual); Study Completion 2012-08 (Actual)

PRIMARY OUTCOMES:
Area under the serum insulin degludec concentration-of s.c. administration | From 0 to infinity after single dose
Area under the serum insulin degludec concentration-of i.v. administration | From 0 to infinity after single dose

SECONDARY OUTCOMES:
Terminal half-life for insulin degludec | From 0 to 30 hours after single dose
Volume of distribution of insulin degludec, estimated during the terminal phase | From 0 to 30 hours after single dose

CONTACTS AND LOCATIONS:
Overall Officials: Global Clinical Registry (GCR, 1452), Study Director — Novo Nordisk A/S
Locations (1):
- Neuss, Germany

REFERENCES:
- See also: Clinical Trials at Novo Nordisk — http://novonordisk-trials.com